CLINICAL TRIAL: NCT03238170
Title: An Exploratory Study to Assess the Feasibility of Incorporating MR in the Radiotherapy Pathway of Patients With Prostate Cancer
Brief Title: MR-simulation in Radiotherapy for Prostate Cancer
Acronym: FIMRA-P
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 215681
Record Dates: First submitted 2017-03-07; First posted 2017-08-03 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Cancer of the PROSTATE
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR-Simulation (Experimental): Patients will have 1 MRI scan appointment, using the Siemens Aera® (Siemens AG Healthcare, Erlangen, Germany) on the same day as their treatment planning CT scan. The MR scan will be performed in the radiotherapy treatment position.
  Interventions: Device: MRI scan

INTERVENTIONS:
Device: MRI scan — MRI scan using the Siemens Aera® (Siemens AG Healthcare, Erlangen, Germany) on the same day as their treatment planning CT scan

SUMMARY:
To assess the feasibility of acquiring an MR scan in the radiotherapy treatment position as part of the patient's radiotherapy pathway and incorporating the data into our radiotherapy planning systems, so that it can be potentially used to reduce healthy tissue exposure to radiation. Subsequently, the protocols and procedures established can be used to put the technique into routine clinical practice.

DETAILED DESCRIPTION:
Conventional radiotherapy treatment planning uses computed tomography (CT) scans to provide an accurate 3-D picture of the local anatomy. This helps the planners to maximise the radiation dose delivered to the prostate, whilst minimising the dose to surrounding normal tissue. Magnetic resonance imaging (MRI) scanning is an established diagnostic imaging technique that provides even clearer images of the local anatomy. However, until recently the technology hasn't existed to allow us to perform MRI scans with patients "set-up" in the position required to plan and deliver radiotherapy to the prostate. This study is being performed to assess methods that may allow us to incorporate MRI scans into the radiotherapy planning process, which may further increase the accuracy of the treatment, reducing the irradiation of surrounding normal tissue and minimising toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Written, voluntary, informed consent
* Age ≥ 18
* ECOG Performance Status ≤ 2
* Life expectancy > 12 months
* Histologically proven carcinoma of the prostate
* Radical radiotherapy +/- hormones indicated as the primary treatment modality
* Staging diagnostic MRI of the prostate need to be available for comparison.
* Adequate organ function and absence of other major concurrent illness, allowing

Exclusion Criteria:

* Inability to provide informed consent
* Impaired renal function (serum creatinine of > 200)
* Severely impaired liver function
* Patients with allergies or contra-indications to the gadolinium contrast agent that may be used in the study
* Severe claustrophobia or inability to tolerate MRI scans
* General contra-indications to MRI including cardiac pacemakers and defibrillators, metallic prosthetic devices, aneurysm clips and metal fragments in the eyes, as defined in MRI safety departmental protocols
* Serious inter-current conditions or other non-malignant illnesses that are uncontrolled or whose control may be affected by participation in this study
* Any patient who has urinary or faecal incontinence
* Status greater than or equal to 3

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Standard Operating Procedure (SOP) for MRI-simulation for prostate patients | 6 months
  Write a Standard Operating Procedure (SOP) for MRI-scanning of prostate patients in the radiotherapy treatment position so that their data can be used in the treatment planning for either in-direct or MRI-only planning

SECONDARY OUTCOMES:
Clinical Protocol for in-direct MRI planning for prostate | 6 months
  Write a clinical protocol for "in-direct" MRI planning of prostate external beam radiotherapy, whereby MRI data is used to define anatomical structures and these are translated onto the co-registered CT scan for treatment planning
Clinical Protocol for direct MRI-only planning for prostate | 18 months
  Write a clinical protocol for "direct" MRI-only planning of prostate external beam radiotherapy, whereby MRI data is used to define anatomical structures and also for dose calculation and setup verification

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hughes, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St. Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas C, Dregely I, Oksuz I, Guerrero Urbano T, Greener T, King AP, Barrington SF. Effect of synthetic CT on dose-derived toxicity predictors for MR-only prostate radiotherapy. BJR Open. 2024 Jun 3;6(1):tzae014. doi: 10.1093/bjro/tzae014. eCollection 2024 Jan. PMID 38948455